CLINICAL TRIAL: NCT00733551
Title: A Randomized, Double-blind, Ascending Dose Trial to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics, of Repeat Doses of Motilin Receptor Agonist GSK962040 in Male and Female Healthy Volunteers
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of Repeat Oral Doses of GSK962040 Administered to Healthy Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOT109681
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Gastroparesis
Keywords: motilin; gastric emptying; GSK962040; oral dose
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects receiving GSK962040 in cohort 1 (Experimental): Eligible subjects will receive repeat oral doses of GSK962040 given as 10 milligrams once daily tablet for 14 days.
  Interventions: Drug: GSK962040; Drug: Placebo
- Subjects receiving GSK962040 in cohort 2 (Experimental): Eligible subjects will receive repeat oral doses of GSK962040 given as 30 milligrams once daily tablet for 14 days.
  Interventions: Drug: GSK962040; Drug: Placebo
- Subjects receiving GSK962040 in cohort 3 (Experimental): Eligible subjects will receive repeat oral doses of GSK962040 given as 100 milligrams once daily tablet for 14 days.
  Interventions: Drug: GSK962040; Drug: Placebo
- Subjects receiving placebo in cohort 1, 2 and 3 (Placebo Comparator): Eligible subjects will receive repeat oral doses of placebo tablets given once daily for 14 days in cohort 1, 2 and 3.
  Interventions: Drug: GSK962040; Drug: Placebo

INTERVENTIONS:
Drug: GSK962040 — GSK962040 tablets will be available in dosing strengths of 1 milligram, 5 milligrams, 25 milligrams given orally, once daily, in the morning, in a fasted state.
Drug: Placebo — Placebo tablets will be given orally, once daily, in the morning, in a fasted state.

SUMMARY:
This study will evaluate the safety, tolerability and exposure of repeat escalating oral doses of GSK962040.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. In any case, liver function tests must be strictly within the normal range at screening.
* Male or female between 18 and 55 years of age, inclusive.
* Non-smoker for at least 6 months based on smoking history.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL is confirmatory.
* Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for at least 4 days following the last dose of study medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication through at least 4 days after the last dose of study medication.
* Body weight > 50 kg and BMI within the range 18.5 - 29.9 kg/m2 (inclusive).
* QTcB or QTcF < 450 msec or QTc<480msec in subjects with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.
* Normal physical examination (physical exam demonstrates no evidence of clinically active disease or physical or mental impairment). A subject with a clinical abnormality may be included only if the Principal Investigator or physician designee considers that the abnormality will not introduce additional risk factors and will not interfere with the study procedures. Consultation with the GSK medical monitor is required before such subjects may be included.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subjects will have negative Helicobacter pylori status or have received eradication within the last calendar year.

Exclusion Inclusion:

* History or presence of any clinically significant metabolic condition, gastrointestinal (including passing of > 3 stools/ day or <3 stools/week) condition or endocrinological condition.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of major gastrointestinal surgical procedure within the last 10 years.
* History of cholecystectomy or biliary tract disease.
* History or presence of thyroid dysfunction (NOTE: subjects with abnormal TSH at screening/baseline or hypothyroidism on a stable dose of thyroid replacement therapy are not eligible).
* A history or presence of recreational drug abuse or dependence or current abuse as evidenced by positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to approximately a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test (from the first urine of the day) at screening or prior to dosing.
* Lactating or pregnant females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* For male volunteers: An unwillingness of the male subject to comply with the contraception requirements listed in the protocol, from the time of the first dose of study medication until at least 4 days following administration of the last dose of study medication.
* History of or current lactose intolerance.
* Subjects recruited for/participating in Cohorts 2-5 will be screened such that subjects exhibiting rapid gastric emptying rates will be excluded, as defined by the reference range of baseline gastric emptying rate (t1/2b) observed in cohort 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09-23 (Actual); Primary Completion 2009-07-20 (Actual); Study Completion 2009-07-20 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and PK of GSK962040 from all adverse event reporting, 12-lead ECGs, vital signs, observation, safety laboratory tests and GI symptom diary; (AUC, Cmax, Tmax, accumulation ratio (Ro), half life and time invariance ratio (Rs)).

SECONDARY OUTCOMES:
Effect on gastric emptying.Effect of liquid meal on PK of GSK962040. Effect on bowel movement parameters
Pharmacokinetic parameters following repeated oral doses of GSK962040 during a simulated liquid enteral feed meal: Cmax, Tmax, and AUC(0-t)
Gastric emptying, as measured by the 13C octanoic acid breath test:Gastric half emptying time (t1/2b), Duration of the lag time (tlag), Gastric evacuation coefficient (GEC)
Bowel movement parameters: Time to first bowel movement after first dose, Daily bowel movement count, Daily average bowel movement Bristol Stool Form scale
Pharmacokinetic parameters following repeated every other day (QOD) oral doses of GSK962040: Cmax, Tmax, AUC(0-t), accumulation ratio (Ro), and, if possible, half-life, and time invariance ratio (Rs), as needed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MOT109681 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MOT109681?search=study&study_ids=109681#rs
- Available data/document: Study Protocol: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MOT109681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register